CLINICAL TRIAL: NCT03765411
Title: Safe Surgery in the Elderly: A Review of Outcomes Following Robotic Proctectomy From the Nationwide Inpatient Sample, a Retrospective Cross Sectional Cohort Study. Cross-Sectional Study
Brief Title: Safe Colorectal Surgery in the Elderly
Status: Completed | Type: Observational
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carly R Richards, General Surgery Chief Resident Surgeon, Tripler Army Medical Center
Other Study IDs: Robotic Proct in the Elderly
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open Proctectomy Patients: Patients who underwent Proctectomy through an open approach
  Interventions: Procedure: Proctectomy
- Laparoscopic Proctectomy Patients: Patients who underwent Proctectomy through a Laparoscopic approach
  Interventions: Procedure: Proctectomy
- Robotic Proctectomy Patients: Patients who underwent Proctectomy through a Robotic approach
  Interventions: Procedure: Proctectomy

INTERVENTIONS:
Procedure: Proctectomy — Resection of the rectum

SUMMARY:
The objective was to evaluate the use and outcomes of robotic proctectomy compared to open and laparoscopic approaches for rectal cancer in the elderly. A retrospective cross-sectional cohort study utilizing the Nationwide Inpatient Sample (NIS; 2006-2013) was performed.

DETAILED DESCRIPTION:
The objective was to evaluate the use and outcomes of robotic proctectomy compared to open and laparoscopic approaches for rectal cancer in the elderly. A retrospective cross-sectional cohort study utilizing the Nationwide Inpatient Sample (NIS; 2006-2013) was performed. All cases were restricted to age 70 years old or greater. The incidence of robotic proctectomy from 2006 - 2013 both as a whole as well as divided into approach was analyzed. Each approach was compared for both primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* underwent proctectomy

Exclusion Criteria:

* emergent admissions
* abdominoperineal resections

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients were eligible if they were 70 years old or greater, underwent proctectomy in an elective setting, and did not have an abdominoperioneal resection.
Sampling Method: Probability Sample
Enrollment: 6740 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
In-hospital Complications | through study completion, an average of 5 days
  Complications to include mechanical wound, infections, urinary, pulmonary, gastrointestinal, cardiovascular, systemic, surgical, and any complication

SECONDARY OUTCOMES:
In-hospital mortality | through study completion, an average of 5 days
  Death during admission
Length of Stay | through study completion, an average of 5 days
  Length of in hospital stay
Costs and Charges | through study completion, an average of 5 days
  Hospital charges refer to the total amount billed by the hospital. Hospital cost refers to the amount paid by the insurance provider

CONTACTS AND LOCATIONS:
Locations (1):
- Tripler Army Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guiding principles for the care of older adults with multimorbidity: an approach for clinicians. Guiding principles for the care of older adults with multimorbidity: an approach for clinicians: American Geriatrics Society Expert Panel on the Care of Older Adults with Multimorbidity. J Am Geriatr Soc. 2012 Oct;60(10):E1-E25. doi: 10.1111/j.1532-5415.2012.04188.x. Epub 2012 Sep 19. No abstract available. PMID 22994865
- [Result] Fielding LP, Phillips RK, Hittinger R. Factors influencing mortality after curative resection for large bowel cancer in elderly patients. Lancet. 1989 Mar 18;1(8638):595-7. doi: 10.1016/s0140-6736(89)91618-8. PMID 2564119
- [Result] Tan KY, Kawamura Y, Mizokami K, Sasaki J, Tsujinaka S, Maeda T, Konishi F. Colorectal surgery in octogenarian patients--outcomes and predictors of morbidity. Int J Colorectal Dis. 2009 Feb;24(2):185-9. doi: 10.1007/s00384-008-0615-9. Epub 2008 Dec 3. PMID 19050901
- [Result] Law WL, Chu KW, Tung PH. Laparoscopic colorectal resection: a safe option for elderly patients. J Am Coll Surg. 2002 Dec;195(6):768-73. doi: 10.1016/s1072-7515(02)01483-7. PMID 12495308
- [Result] Cheung HY, Chung CC, Fung JT, Wong JC, Yau KK, Li MK. Laparoscopic resection for colorectal cancer in octogenarians: results in a decade. Dis Colon Rectum. 2007 Nov;50(11):1905-10. doi: 10.1007/s10350-007-9070-x. Epub 2007 Sep 26. PMID 17899275
- [Result] Stocchi L, Nelson H, Young-Fadok TM, Larson DR, Ilstrup DM. Safety and advantages of laparoscopic vs. open colectomy in the elderly: matched-control study. Dis Colon Rectum. 2000 Mar;43(3):326-32. doi: 10.1007/BF02258297. PMID 10733113
- [Result] Vignali A, Di Palo S, Tamburini A, Radaelli G, Orsenigo E, Staudacher C. Laparoscopic vs. open colectomies in octogenarians: a case-matched control study. Dis Colon Rectum. 2005 Nov;48(11):2070-5. doi: 10.1007/s10350-005-0147-0. PMID 16086219
- [Result] Champagne BJ, Delaney CP. Laparoscopic approaches to rectal cancer. Clin Colon Rectal Surg. 2007 Aug;20(3):237-48. doi: 10.1055/s-2007-984868. PMID 20011205
- [Result] Jayne DG, Brown JM, Thorpe H, Walker J, Quirke P, Guillou PJ. Bladder and sexual function following resection for rectal cancer in a randomized clinical trial of laparoscopic versus open technique. Br J Surg. 2005 Sep;92(9):1124-32. doi: 10.1002/bjs.4989. PMID 15997446
- [Result] van der Pas MH, Haglind E, Cuesta MA, Furst A, Lacy AM, Hop WC, Bonjer HJ; COlorectal cancer Laparoscopic or Open Resection II (COLOR II) Study Group. Laparoscopic versus open surgery for rectal cancer (COLOR II): short-term outcomes of a randomised, phase 3 trial. Lancet Oncol. 2013 Mar;14(3):210-8. doi: 10.1016/S1470-2045(13)70016-0. Epub 2013 Feb 6. PMID 23395398
- [Result] Park S, Kim NK. The Role of Robotic Surgery for Rectal Cancer: Overcoming Technical Challenges in Laparoscopic Surgery by Advanced Techniques. J Korean Med Sci. 2015 Jul;30(7):837-46. doi: 10.3346/jkms.2015.30.7.837. Epub 2015 Jun 10. PMID 26130943
- [Result] Baik SH, Kwon HY, Kim JS, Hur H, Sohn SK, Cho CH, Kim H. Robotic versus laparoscopic low anterior resection of rectal cancer: short-term outcome of a prospective comparative study. Ann Surg Oncol. 2009 Jun;16(6):1480-7. doi: 10.1245/s10434-009-0435-3. Epub 2009 Mar 17. PMID 19290486
- [Result] Kim JY, Kim NK, Lee KY, Hur H, Min BS, Kim JH. A comparative study of voiding and sexual function after total mesorectal excision with autonomic nerve preservation for rectal cancer: laparoscopic versus robotic surgery. Ann Surg Oncol. 2012 Aug;19(8):2485-93. doi: 10.1245/s10434-012-2262-1. Epub 2012 Mar 21. PMID 22434245
- [Result] D'Annibale A, Pernazza G, Monsellato I, Pende V, Lucandri G, Mazzocchi P, Alfano G. Total mesorectal excision: a comparison of oncological and functional outcomes between robotic and laparoscopic surgery for rectal cancer. Surg Endosc. 2013 Jun;27(6):1887-95. doi: 10.1007/s00464-012-2731-4. Epub 2013 Jan 5. PMID 23292566
- [Result] Frasson M, Braga M, Vignali A, Zuliani W, Di Carlo V. Benefits of laparoscopic colorectal resection are more pronounced in elderly patients. Dis Colon Rectum. 2008 Mar;51(3):296-300. doi: 10.1007/s10350-007-9124-0. Epub 2008 Jan 15. PMID 18197453
- [Result] Jayne D, Pigazzi A, Marshall H, Croft J, Corrigan N, Copeland J, Quirke P, West N, Rautio T, Thomassen N, Tilney H, Gudgeon M, Bianchi PP, Edlin R, Hulme C, Brown J. Effect of Robotic-Assisted vs Conventional Laparoscopic Surgery on Risk of Conversion to Open Laparotomy Among Patients Undergoing Resection for Rectal Cancer: The ROLARR Randomized Clinical Trial. JAMA. 2017 Oct 24;318(16):1569-1580. doi: 10.1001/jama.2017.7219. PMID 29067426
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998 Jan;36(1):8-27. doi: 10.1097/00005650-199801000-00004. PMID 9431328
- [Result] Washington CW, Derdeyn CP, Dacey RG Jr, Dhar R, Zipfel GJ. Analysis of subarachnoid hemorrhage using the Nationwide Inpatient Sample: the NIS-SAH Severity Score and Outcome Measure. J Neurosurg. 2014 Aug;121(2):482-9. doi: 10.3171/2014.4.JNS131100. Epub 2014 Jun 20. PMID 24949676
- [Result] Singh JA, Kwoh CK, Boudreau RM, Lee GC, Ibrahim SA. Hospital volume and surgical outcomes after elective hip/knee arthroplasty: a risk-adjusted analysis of a large regional database. Arthritis Rheum. 2011 Aug;63(8):2531-9. doi: 10.1002/art.30390. PMID 21656509
- [Result] Schlussel AT, Lustik MB, Johnson EK, Maykel JA, Champagne BJ, Damle A, Ross HM, Steele SR. A nationwide assessment comparing nonelective open with minimally invasive complex colorectal procedures. Colorectal Dis. 2016 Mar;18(3):301-11. doi: 10.1111/codi.13113. PMID 26362693
- [Result] Damle A, Damle RN, Flahive JM, Schlussel AT, Davids JS, Sturrock PR, Maykel JA, Alavi K. Diffusion of technology: Trends in robotic-assisted colorectal surgery. Am J Surg. 2017 Nov;214(5):820-824. doi: 10.1016/j.amjsurg.2017.03.020. Epub 2017 Mar 21. PMID 28347491
- [Result] Lee MG, Chiu CC, Wang CC, Chang CN, Lee SH, Lee M, Hsu TC, Lee CC. Trends and Outcomes of Surgical Treatment for Colorectal Cancer between 2004 and 2012- an Analysis using National Inpatient Database. Sci Rep. 2017 May 17;7(1):2006. doi: 10.1038/s41598-017-02224-y. PMID 28515452
- [Result] Halabi WJ, Kang CY, Jafari MD, Nguyen VQ, Carmichael JC, Mills S, Stamos MJ, Pigazzi A. Robotic-assisted colorectal surgery in the United States: a nationwide analysis of trends and outcomes. World J Surg. 2013 Dec;37(12):2782-90. doi: 10.1007/s00268-013-2024-7. PMID 23564216
- [Result] Tam MS, Kaoutzanis C, Mullard AJ, Regenbogen SE, Franz MG, Hendren S, Krapohl G, Vandewarker JF, Lampman RM, Cleary RK. A population-based study comparing laparoscopic and robotic outcomes in colorectal surgery. Surg Endosc. 2016 Feb;30(2):455-463. doi: 10.1007/s00464-015-4218-6. Epub 2015 Apr 17. PMID 25894448
- [Result] Baek JH, Pastor C, Pigazzi A. Robotic and laparoscopic total mesorectal excision for rectal cancer: a case-matched study. Surg Endosc. 2011 Feb;25(2):521-5. doi: 10.1007/s00464-010-1204-x. Epub 2010 Jul 7. PMID 20607559
- [Result] Schlussel AT, Delaney CP, Maykel JA, Lustik MB, Nishtala M, Steele SR. A National Database Analysis Comparing the Nationwide Inpatient Sample and American College of Surgeons National Surgical Quality Improvement Program in Laparoscopic vs Open Colectomies: Inherent Variance May Impact Outcomes. Dis Colon Rectum. 2016 Sep;59(9):843-54. doi: 10.1097/DCR.0000000000000642. PMID 27505113
- [Result] Antoniou SA, Antoniou GA, Koch OO, Pointner R, Granderath FA. Laparoscopic colorectal surgery confers lower mortality in the elderly: a systematic review and meta-analysis of 66,483 patients. Surg Endosc. 2015 Feb;29(2):322-33. doi: 10.1007/s00464-014-3672-x. Epub 2014 Jul 2. PMID 24986017
- [Result] Seishima R, Okabayashi K, Hasegawa H, Tsuruta M, Shigeta K, Matsui S, Yamada T, Kitagawa Y. Is laparoscopic colorectal surgery beneficial for elderly patients? A systematic review and meta-analysis. J Gastrointest Surg. 2015 Apr;19(4):756-65. doi: 10.1007/s11605-015-2748-9. Epub 2015 Jan 24. PMID 25617077
- [Result] Park JS, Choi GS, Lim KH, Jang YS, Jun SH. Robotic-assisted versus laparoscopic surgery for low rectal cancer: case-matched analysis of short-term outcomes. Ann Surg Oncol. 2010 Dec;17(12):3195-202. doi: 10.1245/s10434-010-1162-5. Epub 2010 Jun 30. PMID 20589436
- [Result] Keller DS, Senagore AJ, Lawrence JK, Champagne BJ, Delaney CP. Comparative effectiveness of laparoscopic versus robot-assisted colorectal resection. Surg Endosc. 2014 Jan;28(1):212-21. doi: 10.1007/s00464-013-3163-5. Epub 2013 Aug 31. PMID 23996335
- [Result] Li Y, Wang S, Gao S, Yang C, Yang W, Guo S. Laparoscopic colorectal resection versus open colorectal resection in octogenarians: a systematic review and meta-analysis of safety and efficacy. Tech Coloproctol. 2016 Mar;20(3):153-62. doi: 10.1007/s10151-015-1419-x. Epub 2016 Jan 18. PMID 26783029
- [Result] Park JS, Choi GS, Lim KH, Jang YS, Jun SH. S052: a comparison of robot-assisted, laparoscopic, and open surgery in the treatment of rectal cancer. Surg Endosc. 2011 Jan;25(1):240-8. doi: 10.1007/s00464-010-1166-z. Epub 2010 Jun 15. PMID 20552367
- [Result] Agha RA, Borrelli MR, Vella-Baldacchino M, Thavayogan R, Orgill DP; STROCSS Group. The STROCSS statement: Strengthening the Reporting of Cohort Studies in Surgery. Int J Surg. 2017 Oct;46:198-202. doi: 10.1016/j.ijsu.2017.08.586. Epub 2017 Sep 7. PMID 28890409
- See also: An Aging World: 2015 International Population Reports — https://www.census.gov/content/dam/Census/library/publications/2016/demo/p95-16-1.pdf
- See also: Overview of the Nationwide Inpatient Sample. [Internet].; 2017 — http://www.hcup-us.ahrq.gov/nisoverview.jsp
- See also: All patient refined diagnosis related groups (APR-DRGs), version 20.0. methodology overview — http://www.hcup-us.ahrq.gov/db/nation/nis/APR-DRGsV20MethodologyOverviewandBibliography.pdf